CLINICAL TRIAL: NCT03459196
Title: Clinical Study for Safety and Acute Performance Evaluation of the THERMOCOOL SMARTTOUCH® SF-5D System Used With Fast Ablation Mode in Treatment of Patients With Paroxysmal Atrial Fibrillation.
Acronym: QDOT-FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI_2017_02
Record Dates: First submitted 2018-02-23; First posted 2018-03-08 (Actual); Results first posted 2019-11-06 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Interventional; Radiofrequency Ablation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): A novel radiofrequency ablation catheter combining microelectrodes, thermocouples, porous tip irrigation and contact force sensing nMARQ Multi-Channel RF Generator with Software including TGA mode (Temperature Guided Ablation).
  Interventions: Device: THERMOCOOL SMARTTOUCH SF-5D Catheter

INTERVENTIONS:
Device: THERMOCOOL SMARTTOUCH SF-5D Catheter — radiofrequence ablation with THERMOCOOL SMARTTOUCH® SF-5D catheter used in combination with the nMARQ™ Multi-Channel RF Generator with TGA mode

SUMMARY:
The QDOT-FAST study is a prospective, multi-center, non-randomized, interventional clinical study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate safety and acute performance of the THERMOCOOL SMARTTOUCH® SF-5D catheter used in combination with the nMARQ™ Multi-Channel RF Generator with TGA mode in the treatment of Paroxysmal Atrial Fibrillation (PAF) during standard electrophysiology mapping and RF ablation procedures.

The QDOT-FAST study is a prospective, multi-center, non-randomized, interventional clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Signed the Patient Informed Consent Form (ICF).
3. Diagnosed with symptomatic PAF
4. Selected for catheter ablation through pulmonary vein isolation.
5. Able and willing to comply with all pre-, post-, and follow-up testing and requirements (e.g. patient not confined by a court ruling).

Exclusion Criteria:

1. Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
2. Previous surgical or catheter ablation for atrial fibrillation.
3. Previously diagnosed with persistent, longstanding AF and/or continuous AF >7 days, or >48 hrs. terminated by cardioversion.
4. Documented Left Atrial thrombus on baseline/pre-procedure imaging.
5. Any carotid stenting or endarterectomy.
6. Left atrial (LA) size >50mm.
7. Left Ventricular ejection fraction (LVEF) <40%.
8. Uncontrolled heart failure or New York Heart Association (NYHA) function class III or IV.
9. History of blood clotting or bleeding abnormalities
10. Contraindication to anticoagulation
11. History of a documented thromboembolic event (including transient ischemic attack (TIA)) within the past 12 months.
12. Previous percutaneous coronary intervention (PCI) or myocardial Infarction (MI) within the past 2 months.
13. Coronary artery bypass grafting (CABG) in conjunction with valvular surgery, cardiac surgery (e.g. ventriculotomy, atriotomy) or valvular cardiac (surgical or percutaneous) procedure.
14. Rheumatic Heart Disease
15. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months.
16. Unstable angina.
17. Significant pulmonary disease (e.g. restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other diseaseor malfunction of the lungs or respiratory system that produces chronic symptoms.
18. Acute illness, active systemic infection, or sepsis.
19. Presence of atrial myxoma, interatrial baffle or patch
20. Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction or manipulation.
21. Presence of a condition that precludes vascular access.
22. Presence of implanted pacemaker or implantable cardioverter-defibrillator (ICD).
23. Presence of IVC filter
24. Significant congenital anomaly or a medical problem that in the opinion of the investigator would preclude enrollment in this trial.
25. Currently enrolled in an investigational study evaluating another device, biologic, or drug.
26. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal), lactating, or who are of child bearing age and plan on becoming pregnant during the course of the clinical investigation.
27. Life expectancy or other disease processes likely to limit survival to less than 12 months.
28. Presenting contra-indication for the devices used in the study, as indicated in the respective instructions for use.
29. Categorized as vulnerable population and requires special treatment with respect to safeguards of well-being
30. Contraindication to use of contrast agents for MRI such as advanced renal disease, etc. (at PI discretion)
31. Presence of iron-containing metal fragments in the body
32. Unresolved pre-existing neurological deficit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Elisabethinen Hospital, Linz, Austria
- Belgium (3):
  - OLV Aalst, Aalst
  - AZ Sint-Jan, Bruges
  - Jessa Ziekenhuis, Hasselt
- Czechia (2):
  - Ceské Budejovice Hospital, České Budějovice
  - Na Homolce, Prague
- Ospedale F Miulli, Bari, Italy

REFERENCES:
- [Derived] Reddy VY, Grimaldi M, De Potter T, Vijgen JM, Bulava A, Duytschaever MF, Martinek M, Natale A, Knecht S, Neuzil P, Purerfellner H. Pulmonary Vein Isolation With Very High Power, Short Duration, Temperature-Controlled Lesions: The QDOT-FAST Trial. JACC Clin Electrophysiol. 2019 Jul;5(7):778-786. doi: 10.1016/j.jacep.2019.04.009. Epub 2019 May 8. PMID 31320006
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=BWI_2017_02&attachmentIdentifier=e7466843-5acf-4d13-aa3f-9b175af83913&fileName=1_Appendix_A_Protocol_v1.0_21Dec2017_Redacted_7Aug2019.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 54 subjects were enrolled in the study at 7 sites in Europe. The first subject was enrolled on April 17th, 2018 and the last subject was enrolled on June 20th, 2018.
Pre-assignment Details: Subjects were screened carefully prior to enrollment in the study to ensure compliance with the inclusion and exclusion criteria. All subjects were screened using pre-procedure imaging for the presence of LA thrombus, which was intended to decrease the potential for thromboembolic complications.
Groups:
- THERMOCOOL SMARTTOUCH SF-5D Catheter: A novel radiofrequency ablation catheter combining microelectrodes, thermocouples, porous tip irrigation and contact force sensing nMARQ Multi-Channel RF Generator with Software including temperature guided ablation mode.
Period: Overall Study
Arm/Group | THERMOCOOL SMARTTOUCH SF-5D Catheter
Started (Subjects who signed the informed consent form are considered as enrolled and started the study.) | 54
Completed | 52
Not Completed | 2
Not completed — Subject didn't receive study catheter | 2

BASELINE CHARACTERISTICS:
Arm/Group | THERMOCOOL SMARTTOUCH SF-5D Catheter
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  European Union | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieved Acute Procedural Success
Description: Defined acute procedural success as confirmation of entrance block in all targeted pulmonary veins after adenosine or isoproterenol challenge.
Time Frame: Day 1
Population: Effectiveness population includes all subjects who have had the investigational device inserted and underwent ablation with the study catheter used in conjunction with QMode+ for pulmonary vein isolation (PVI). Subjects without any QMode+ application for PVI are excluded from the effectiveness population.
Measure: Count of Participants; unit: Participants
Arm/Group | THERMOCOOL SMARTTOUCH SF-5D Catheter
Number analyzed (Participants) | 52
Participants | 52

2. Primary Outcome: Incidence of Acute Safety
Description: Defined as the incidence of early-onset predefined primary adverse events within 7 days of the study procedure, including atrio-eophageal fistula, phrenic nerve paralysis , cardiac tamponade/perforation , pulmonary vein stenosis, death, stroke/CVA, major vascular access complication/bleeding , thromboembolism, myocardial infarction, transient ischemic attack. Device or procedure related death, pulmonary vein stenosis and atrio-esophageal fistula that occur beyond 7 days post- procedure were also be deemed primary AEs.
Time Frame: 7 days post-procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | THERMOCOOL SMARTTOUCH SF-5D Catheter
Number analyzed (Participants) | 52
Participants | 2

ADVERSE EVENTS:
Time Frame: 3 months post-procedure
Arm/Group | THERMOCOOL SMARTTOUCH SF-5D Catheter
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 4/52
Other Adverse Events (participants affected / at risk) | 32/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL SMARTTOUCH SF-5D Catheter (N=52)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL SMARTTOUCH SF-5D Catheter (N=52)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Diverticulum gastric (Gastrointestinal disorders) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 3 (3)
Gastric disorder (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6)
Hiatus hernia (Gastrointestinal disorders) | 2 (2)
Oesophageal disorder (Gastrointestinal disorders) | 1 (1)
Oesophageal mucosa erythema (Gastrointestinal disorders) | 1 (1)
Oesophageal polyp (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Haematoma (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT03459196/Prot_001.pdf
  • Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT03459196/SAP_000.pdf